CLINICAL TRIAL: NCT02620800
Title: An Open Label, Multicenter, Single Arm, Phase 1/2 Trial of Metronomic 5-fluorouracil in Combination With Nab-paclitaxel, Bevacizumab, Leucovorin, and Oxaliplatin in Patients With Metastatic Pancreatic Adenocarcinoma.
Brief Title: Study of 5-fluorouracil (5-FU), Nab®1-paclitaxel, Bevacizumab, Leucovorin, and Oxaliplatin in Patients With Metastatic Pancreatic Cancer
Acronym: FABLOx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-PANC-009
Record Dates: First submitted 2015-11-30; First posted 2015-12-03 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Pancreas Adenocarcinoma
Keywords: Metastatic Pancreatic Cancer; Adenocarcinoma; Open-label; Phase 1/2; Metronomic; Chemotherapy; ABI-007; nab-paclitaxel; Abraxane; gemcitabine; Gemzar; bevacizumab; Avastin; 5-Fluorouracil (5-FU); leucovorin; oxaliplatin; Eloxatin
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Fluorouracil; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Bevacizumab; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FABLOx (Experimental): 5 fluorouracil (5-FU ) (180 mg/m^2/day for 14 days), by continuous intravenous infusion (CIVI) via ambulatory pump, nab-paclitaxel (75 mg/m^2) as a 30-minute (min) IV infusion on Days 1, 8, and 15, bevacizumab (5 mg/kg) as an IV infusion on Days 1 and 15, calcium leucovorin (20 mg/m^2) IV bolus on Days 1, 8, 15, and oxaliplatin (40 mg/m^2) as a 60-min IV infusion on Days 1, 8, and 15. First bevacizumab infusion is given over 90 minutes.
  Interventions: Drug: 5FU; Drug: nab-paclitaxel; Drug: bevacizumab; Drug: calcium leucovorin; Drug: oxaliplatin

INTERVENTIONS:
Drug: 5FU — 5 fluorouracil (5-FU) (180 mg/m^2/day for 14 days) by CIVI via ambulatory pump
Drug: nab-paclitaxel — nab-paclitaxel (75 mg/m^2) as a 30-minute (min) IV infusion on Days 1, 8, and 15
  Other Names: Abraxane; ABI-007
Drug: bevacizumab — bevacizumab (5 mg/kg) as an IV infusion on Days 1 and 15
  Other Names: Avastin
Drug: calcium leucovorin — calcium leucovorin (20 mg/m^2) IV bolus, on Days 1, 8, 15
  Other Names: Citrovorum Factor; Folinic Acid
Drug: oxaliplatin — oxaliplatin (40 mg/m^2) as a 60-min IV infusion on Days 1, 8, and 15
  Other Names: Elotaxin

SUMMARY:
The purpose of this study is to learn about the safety and potential benefit of metronomic 5-fluorouracil in combination with nab®1-paclitaxel, bevacizumab, leucovorin, and oxaliplatin in treating patients with metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
The Phase 1 portion of the study is an open-label study enrolling subjects with metastatic pancreatic adenocarcinoma who have not previously received systemic chemotherapy at any time as treatment for pancreatic cancer (including adjuvant chemotherapy), except low dose chemotherapy administered as a radiosensitizer concomitant with radiotherapy and to determine the recommended Phase 2 dose (RP2D) and dose-limiting toxicities (DLTs) of metronomic 5-FU in combination with nab-paclitaxel, bevacizumab, leucovorin, and oxaliplatin in patients with metastatic pancreatic adenocarcinoma.

Subjects will be enrolled in cohorts of 6 subjects. There will be no dose escalation. Dose limiting toxicities will be assessed in cycle 1. If there is an incidence of ≥2 of 6 subjects experiencing a DLT, the dose will be de-escalated to the next lower dose. Based on the totality of the data, the investigators may advise the Sponsor to evaluate additional subjects at any of the dose levels. Upon Sponsor agreement, if additional subjects are enrolled at any dose level, DLT evaluation will occur at that same ratio (if ≥ 4 of 12 subjects, or ≥ 6 of 18 subjects experience a DLT, the dose will be de-escalated). Approximately 12-24 subjects will be enrolled in the Phase 1 portion of the study, dependent on the number of dose levels examined and the number of subjects enrolled at each dose level.

Safety will continuously be evaluated by incidence of Treatment Emergent Adverse Events (TEAEs) by the Medical Dictionary for Drug Regulatory Activities (MedDRA) and severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 (v4.03).

The Phase 2 part of the study is to determine if the combination of metronomic 5-FU, nab-paclitaxel, bevacizumab, leucovorin, and oxaliplatin at the RP2D defined in Phase 1 achieves a clinically meaningful improvement in 1 year survival rate over the historical control. Approximately 60 subjects are planned to be enrolled in the Phase 2 portion of the study.

Subjects may remain on treatment until disease progression, unacceptable toxicity, withdrawal of consent, physician decision, or death. The anticipated duration of the study (including Phase 1, Phase 2 and follow-up) is approximately 4 years.

The Phase 1 portion of the study is an open-label study enrolling subjects with metastatic pancreatic adenocarcinoma who have not previously received systemic chemotherapy at any time as treatment for pancreatic cancer (including adjuvant chemotherapy), except low dose chemotherapy administered as a radiosensitizer concomitant with radiotherapy and to determine the recommended Phase 2 dose (RP2D) and dose-limiting toxicities (DLTs) of metronomic 5-FU in combination with nab-paclitaxel, bevacizumab, leucovorin, and oxaliplatin in patients with metastatic pancreatic adenocarcinoma.

Subjects will be enrolled in cohorts of 6 subjects. There will be no dose escalation. Dose limiting toxicities will be assessed in cycle 1. If there is an incidence of ≥2 of 6 subjects experiencing a DLT, the dose will be de-escalated to the next lower dose. Based on the totality of the data, the investigators may advise the Sponsor to evaluate additional subjects at any of the dose levels. Upon Sponsor agreement, if additional subjects are enrolled at any dose level, DLT evaluation will occur at that same ratio (if ≥ 4 of 12 subjects, or ≥ 6 of 18 subjects experience a DLT, the dose will be de-escalated). Approximately 12-24 subjects will be enrolled in the Phase 1 portion of the study, dependent on the number of dose levels examined and the number of subjects enrolled at each dose level.

Safety will continuously be evaluated by incidence of Treatment Emergent Adverse Events (TEAEs) by the Medical Dictionary for Drug Regulatory Activities (MedDRA) and severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 (v4.03).

The Phase 2 part of the study is to determine if the combination of metronomic 5-FU, nab-paclitaxel, bevacizumab, leucovorin, and oxaliplatin at the RP2D defined in Phase 1 achieves a clinically meaningful improvement in 1 year survival rate over the historical control. Approximately 60 subjects are planned to be enrolled in the Phase 2 portion of the study.

Subjects may remain on treatment until disease progression, unacceptable toxicity, withdrawal of consent, physician decision, or death. The anticipated duration of the study (including Phase 1, Phase 2 and follow-up) is approximately 4 years.

Upon completion of the Phase 1 portion of the study, a decision not to proceed with the Phase 2 portion was taken by the Sponsor. The decision to terminate the study after Phase 1 was not based on any safety concerns that posed an unacceptable risk for this patient population and no safety issues have been identified.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria are met:

1. Male or female subject is between 18 and 65 years of age at the time of signing the Informed Consent Form (ICF).
2. Subject has definitive histologically or cytologically confirmed metastatic pancreatic adenocarcinoma.
3. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
4. Subject has one or more tumors measurable by CT scan (or (MRI), if allergic to CT contrast media) as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
5. Subject has the following blood counts / Hemoglobin (Hgb) at screening:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   * Platelet count ≥ 100,000/mm3 (100 × 10^9/L);
   * Hgb ≥ LLN or 10 g/dL.
6. Subject has the following blood chemistry levels at screening:

   * AST (SGOT), ALT (SGPT) ≤ 2.5 x upper limit of normal range (ULN); if hepatic metastases present ≤ 5.0 x ULN
   * Total bilirubin ≤ 1.5 X ULN
   * Creatinine clearance ≥ 60 mL/min (by Cockroft-Gault)
   * Albumin ≥ 3.5 grams/dL7.
7. Females of childbearing potential (FOCBP) [defined as a sexually mature woman who (1) have not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months)] must:

   * Have a negative pregnancy test (β-human chorionic gonadotropin [β -hCG]) as verified by the study doctor within 72 hours prior to starting study therapy
   * Commit to complete abstinence from heterosexual contact, or agree to use medical doctor-approved contraception throughout the study without interruption; while receiving study medication and for at least 6 months following last dose of study IP.
8. Males must practice complete abstinence or agree to use a condom (even if he has undergone a successful vasectomy) during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 6 months following last dose of study IP.
9. Subject has no clinically significant abnormalities in urinalysis results at baseline.
10. Subject is able to adhere to the study visit schedule and other protocol requirements.
11. Subject understands the nature of the study, and has agreed to participate in the study, and has voluntarily signed the ICF prior to participation in any study-related activities.
12. Subject must consent to provide protocol-mandated tumor and blood samples for molecular analysis.
13. Subject is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Subject has received previous systemic chemotherapy or investigational therapy (other than that as a radiosensitizer concomitant with radiotherapy) for the treatment of pancreatic adenocarcinoma, including neo-adjuvant or adjuvant therapy.
2. Subject has known brain metastases unless previously treated and controlled for a minimum of 2 weeks prior to enrollment. Subject is not receiving corticosteroids with no evidence of cerebral edema.
3. Pre-existing peripheral neuropathy > Grade 1
4. Subject with unstable stent.
5. History of malignancy in the last 3 years. Subjects with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Subjects with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 3 years.
6. Subject has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy , defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
7. Subject has known historical or active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C or subject receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the Investigator, increase the risk of serious neutropenic complications.
8. Subject has undergone major surgery, other than diagnostic surgery (ie, surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study or surgical wound has not fully healed.
9. Subject has a history of allergy or hypersensitivity to any of the IP or any of their excipients, or the subject exhibits any of the events outlined in the Contraindications or Special Warnings and Precautions sections for and of the products' Summary of Product Characteristics or Prescribing Information.
10. History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa).
11. Subject with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies that in the opinion of the Investigator may put them at increased risk of interstitial pneumonitis.
12. Subject with high cardiovascular risk, including, but not limited to:

    * uncontrolled hypertension
    * unstable angina
    * diagnosis of ischemic heart disease
    * heart disease of New York Heart Association functional classification ≥ 3 (see Appendix C)
    * prior history of hemorrhagic or thrombolytic stroke
    * prior exposure to anthracycline
    * history of peripheral artery disease (eg, claudication, Leo Buerger's disease)
    * any of the following within the prior 6 months
    * coronary stenting
    * myocardial infarction
    * coronary bypass surgery
13. Recent history of clinically significant hemoptysis.
14. Pregnant and nursing (lactating) women.
15. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
16. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
17. Subject has any condition that confounds the ability to interpret data from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (Phase 1) | Up to Day 1 of Cycle 2
  • Any toxicity starting during the first 28 days of treatment and requiring 14 days or more of treatment interruption • Grade 3 or 4 neutropenia associated with fever > 38.5°C • Grade 3 anemia requiring a transfusion • Any Grade 4 hematological toxicity lasting > 7 days • Grade 4 thrombocytopenia or a Grade 3 or 4 thrombocytopenia associated with clinically significant bleeding • Grade 3 or 4 non-hematological toxicity with the exception of fatigue, due to any of the study drugs and unresponsive to medical treatment within 4 days of onset • Subjects who experience Grade ≥ 3 hyperbilirubinemia as an apparent DLT. If a Phase 1 subject experiences a Grade ≥ 3 hyperbilirubinemia due principally to unconjugated bilirubin, it will not be defined as a DLT. The subject will be removed from the study and the Phase 1 subject will be replaced. • Any non-hematologic toxicity delaying the initiation of cycle 2 by > 21 days • Grade ≥ 2 pneumonitis or interstitial lung disease
1 year survival rate (Phase II portion) | Up to 1 year
  1 year survival rate is defined as the time interval between the date of first dose of Investigational Product (IP) and the date of death.
Number of subjects experiencing Adverse Events (AEs) by severity and overall tabulations by cohort and overall including treatment emergent and Serious AEs | Up to 4 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. All AEs will be recorded by the Investigator from the time the subject signs informed consent until 28 days after the last dose of IP as well as those SAEs made known to the Investigator at any time thereafter that are suspected of being related to Investigational Product.

SECONDARY OUTCOMES:
Summary for the number of subjects experiencing Adverse Events (AEs) by severity and overall in tabulations by cohort and overall including treatment emergent AEs and Serious AEs | Up to 4 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. All AEs will be recorded by the Investigator from the time the subject signs informed consent until 28 days after the last dose of IP as well as those SAEs made known to the Investigator at any time thereafter that are suspected of being related to IP
Objective Response Rate using Response Evaluation Criteria In Solid Tumours (Recist) v1.1 presented by frequency and percentages | Up to 4 years
  Subjects with confirmed complete or partial response (CR and PR) will be presented by 95% Confidence Intervals (CIs) around the proportion of (CR+PR)/N where N is the total number of subjects who are evaluable for response by RECIST criteria.
Progression free survival (PFS) | Up to 4 years
  The time interval between the date of first dose of IP until disease progression or death, whichever occurs first.
Overall Survival (OS) | Up to 4 years
  OS is defined as the time interval between the date of first dose of IP and the date of death.
Percentage of subjects with symptom improvement | Up to 4 years
  The Pancreatic cancer symptom management using: Functional Assessment Solid Tumors Hepatobiliary Symptom Index-8 (FHSI-8) questionaire will evaluate individual symptom improvement from baseline will be analyzed by different levels of improvement separately, ie, by reduction of score 1, 2, 3, and 4. At any given follow-up time point, the subject is classified having symptom improvement if the subject has reduced symptom severity compared to baseline regardless of subsequent symptom score.
Percentage of subjects with symptom improvement between subjects who experienced at least partial response and those without partial response | Up to 4 years
  The FHSI-8 assessment will measure the correlation of symptom improvement between those who experienced a Partial Response (PR) to those without a PR.
Percentage of subjects who experienced symptom improvement by a score of ≥ 2 | Up to 4 years
  The FHSI-8 assessment will measure the correlation of symptom improvement with Eastern Cooperative Oncology Group (ECOG) performance status (PS) over the course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chrystal Louis, MD, Study Director — Celgene
Locations (7):
- United States (7):
  - Northwestern University, Chicago, Illinois
  - Tufts - New England Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Center Wayne State University, Detroit, Michigan
  - Cornell University Weill Medical College, New York, New York
  - Gibbs Cancer Center and Research Institute, Spartanburg, South Carolina
  - Virginia Mason Cancer Center, Seattle, Washington